CLINICAL TRIAL: NCT05056025
Title: A PILOT STUDY TO EVALUATE THE PROGRESSION OF THE DISEASE AND RESPONSE TO SUPPLEMENTATION WITH POSTBIOTICS IGEN-0222 IN PATIENTS WITH MACULAR DEGENERATION
Brief Title: Study to Evaluate the Response to Supplementation With Postbiotics in Patients With Macular Degeneration.
Acronym: REVERS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de la Macula y la Retina (Other)
Collaborators: Igen BioLab SLU (Industry)
Responsible Party: Principal Investigator, Jordi Mones MD PhD, Jordi Mones MD, PhD, Institut de la Macula y la Retina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020/79-MIN-HUGC
Record Dates: First submitted 2021-04-15; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: AMD; Soft Drusen; Reticular Pseudodrusen; Drusen Stage Macular Degeneration; Drusen (Degenerative) of Macula, Bilateral
Keywords: postbiotic; vitamins; drusen; intermediate AMD
MeSH Terms: interventions — Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postbiotics with vitamins (Experimental): postbiotics (IGENH35.3A) with vitamins (AREDS formulation and recommended daily dose)
  Interventions: Dietary Supplement: Postbotics and Vitamins
- vitamins (Placebo Comparator): vitamins (AREDS formulation and recommended daily dose)
  Interventions: Dietary Supplement: Vitamins

INTERVENTIONS:
Dietary Supplement: Postbotics and Vitamins — 2 capsule 3 times a day, before meals
  Arms: postbiotics with vitamins
Dietary Supplement: Vitamins — 2 capsule 3 times a day, before meals
  Arms: vitamins

SUMMARY:
A pilot study to establish the efficacy and safety of supplementation with postbiotics in patients with macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged 50 years or older with high risk intermediate AMD defined as the following criteria:

>4 areas of at least iRORA or iORA (incomplete RPE and outer retinal atrophy and incomplete outer retinal atrophy).

1 area of cRORA + 2 > areas of iRORA. < 1 mm2 of cRORA (complete RPE and outer retinal atrophy). No exudative neovascular AMD.

Exclusion Criteria:

Best corrected visual acuity in the study eye less than 20/400 by ETDRS. Not ability to provide written informed consent. Not ability to return for all trial visits. if subject cannot attend all trial required visits. GA secondary to any condition other than specified. Any ocular condition in the study eye that would progress during the study that could affect central vision or otherwise be a confounding factor.

Concomitant treatment with any ocular or systemic medication that is known to be toxic to the lens, retina or optic nerve. Anti -VEGF therapy is allowed in Cohort B.

Presence of intraocular inflammation (≥ trace cell or flare), macular hole, pathologic myopia, epiretinal membrane, evidence of significant vitreo-retinal traction maculopathy, vitreous hemorrhage or aphakia (pseudophakia with or without an intact capsule is not an exclusion criteria).

Presence of idiopathic or autoimmune-associated uveitis in either eye. Significant media opacities, including cataract, which might interfere with visual acuity, assessment of toxicity, fundus photography or fundus autofluorescence. Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the following year.

Any intraocular surgery or thermal laser within three (3) months of trial entry.

Any prior thermal laser in the macular region, regardless of indication. History of any of the following procedures: Posterior vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant or retinal detachment.

Previous therapeutic radiation in the region of the study eye. Any treatment with an investigational agent in the past 60 days for any condition.

Pregnant or nursing women. Additionally, women with childbearing potential must be using at least two effective contraception methods.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Microperimetry | 12 months
  Median change difference in the % reduced threshold in microperimetry
Color vision change | 12 months
  Median change in red/green and yellow/blue color thresholds

SECONDARY OUTCOMES:
Average Threshold microperimetry | 12 months
  Mean change of Average Threshold microperimetry
Best corrected visual acuity (BCVA) | 12 months
  Mean Change of Best corrected visual acuity (BCVA)
Low luminance visual acuity (LLVA) | 12 months
  Mean Change of Low luminance visual acuity (LLVA)
Rod and cone sensitivity | 12 months
  Mean change of Rod and cone sensitivity test
Advanced Vision and Optometric Test (AVOT) | 12 months
  Mean change AVOT vision test
incomplete retinal pigment epithelial and outer retinal atrophy (iRORA) conversion loci | 12 months
  Number of scans within the optical coherence tomography OCT cube as as per protocol (Spectralis OCT cube protocol: 20º x 20ª, 97b-scan, high-resolution, 62 microns between scans centered at the fovea) with features of iRORA2 conversion loci (change from baseline to 12 months of iRORA loci).
complete retinal pigment epithelial and outer retinal atrophy (cRORA) conversion loci | 12 months
  Number of scans within the OCT cube as as per protocol with of features of cRORA (change from baseline to 12 months of cRORA loci).
Area of cumulative cRORA conversion | 12 months
  Area of cumulative cRORA conversion as measured in mm2 by en face OCT projection scans of the OCT cube as as per protocol
Hyperreflective dots(HRD)+ (retinal pigment epithelium)RPE defects areas conversion | 12 months
  Number of scans within the OCT cube as as per protocol with HRD+RPE defects areas conversion (change from baseline to 12 months of HRD+RPE defects)
Change in outer nuclear layer (ONL) volume | 12 months
  Change in outer nuclear layer (ONL) volume measured by the spectralis software after manually correction of the layer segmentation
Change of drusen > 100 microns height | 12 months
  Change of number of drusen of > 100 microns height measured by OCT within the OCT cube as as per protocol
Change of subretinal drusenoid deposits (SDD) through ellipsoid zone (ELZ) | 12 months
  Change of number of subretinal drusenoid deposits (SDD) through ellipsoid zone within the OCT cube as as per protocol
Change of SDD ribbon | 12 months
  Change of number SDD ribbon within the OCT cube as as per protocol
Conversion to choroidal neovascularization (CNV) | 12 months
  Any conversion to any type of macular neovascularization (MNV) within the OCT cube as as per protocol 1 as per OCT features of leakage, and/or intrarretinal, subretinal or subRPE fluid, and/or presence of Subretinal hyperreflective material(SHRM)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Mones, MD, PhD, Principal Investigator — Institut de la Macula
Locations (1):
- Institut de la Macula, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No